CLINICAL TRIAL: NCT03916185
Title: Randomized Phase I/II Study of the Safety and Immunogenicity of a Single Dose of the Recombinant Live-Attenuated Respiratory Syncytial Virus (RSV) Vaccines RSV ΔNS2/Δ1313/I1314L, RSV 6120/ΔNS2/1030s, RSV 276 or Placebo, Delivered as Nose Drops to RSV-Seronegative Children 6 to 24 Months of Age
Brief Title: Safety and Immunogenicity of a Single Dose of the Recombinant Live-Attenuated Respiratory Syncytial Virus (RSV) Vaccines RSV ΔNS2/Δ1313/I1314L, RSV 6120/ΔNS2/1030s, RSV 276 or Placebo, Delivered as Nose Drops to RSV-Seronegative Children 6 to 24 Months of Age
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study closed to enrollment prior to fully accruing due to difficulties with slower than expected accrual.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IMPAACT 2021; 38530 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2019-04-10; First posted 2019-04-16 (Actual); Results first posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-01

CONDITIONS: Respiratory Syncytial Virus (RSV)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- RSV ΔNS2/Δ1313/I1314L Vaccine (Experimental): Participants received a single dose of the RSV ΔNS2/Δ1313/I1314L vaccine at study entry (Day 0).
  Interventions: Biological: RSV ΔNS2/Δ1313/I1314L Vaccine
- RSV 6120/ΔNS2/1030s Vaccine (Experimental): Participants received a single dose of the RSV 6120/ΔNS2/1030s vaccine at study entry (Day 0).
  Interventions: Biological: RSV 6120/ΔNS2/1030s Vaccine
- RSV 276 Vaccine (Experimental): Participants received a single dose of the RSV 276 vaccine at study entry (Day 0).
  Interventions: Biological: RSV 276 Vaccine
- Placebo (Placebo Comparator): Participants received a single dose of placebo at study entry (Day 0).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: RSV ΔNS2/Δ1313/I1314L Vaccine — 10^6 plaque-forming units (PFU); administered as nose drops
  Arms: RSV ΔNS2/Δ1313/I1314L Vaccine
Biological: RSV 6120/ΔNS2/1030s Vaccine — 10^5 plaque-forming units (PFU); administered as nose drops
  Arms: RSV 6120/ΔNS2/1030s Vaccine
Biological: RSV 276 Vaccine — 10^5 plaque-forming units (PFU); administered as nose drops
  Arms: RSV 276 Vaccine
Biological: Placebo — Administered as nose drops
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate the safety and immunogenicity of a single dose of the recombinant live-attenuated respiratory syncytial virus (RSV) vaccines, RSV ΔNS2/Δ1313/I1314L, RSV 6120/ΔNS2/1030s, and RSV 276, in RSV-seronegative children 6 to 24 months of age.

DETAILED DESCRIPTION:
This study evaluated the safety and immunogenicity of a single dose of the recombinant live-attenuated respiratory syncytial virus (RSV) vaccines, RSV ΔNS2/Δ1313/I1314L, RSV 6120/ΔNS2/1030s, and RSV 276, in RSV-seronegative children 6 to 24 months of age.

Participants were randomly assigned to receive a single dose of RSV ΔNS2/Δ1313/I1314L vaccine, RSV 6120/ΔNS2/1030s vaccine, RSV 276 vaccine, or placebo intranasally at study entry.

Participants were enrolled in the study outside of RSV season. All participants were to remain on study until they completed the post-RSV season visit in the calendar year following enrollment. Participants' total study duration was expected to be between 5 and 15 months, depending on when they enrolled in the study and accommodations given for the COVID pandemic.

Participants attended several study visits throughout the study, which included physical examinations, blood collection, and nasal washes or swabs, if applicable. Participants' parents or guardians were contacted by study staff at various times during the study to monitor participants' health.

The study closed to enrollment prior to fully accruing due to difficulties with slower than expected accrual.

ELIGIBILITY:
Inclusion Criteria:

* In good health based on review of the medical record, history, and physical examination, without evidence of chronic disease.
* Parent/guardian is willing and able to provide written informed consent as described in the study protocol.
* Seronegative for RSV antibody, defined as a serum RSV-neutralizing antibody titer less than 1:40 at screening from a sample collected no more than 42 days prior to study product administration.

  * Note: results from specimens collected during screening for any study of an RSV vaccine developed by the Laboratory of Infectious Diseases (LID) (National Institute of Allergy and Infectious Diseases [NIAID], National Institutes of Health [NIH]) are acceptable. If study product will not be administered the same day as randomization (see the study protocol), it must be administered no more than 42 days after the screening sample is collected.
* Growing normally for age in the opinion of the site clinician in the six months prior to enrollment AND has a current height and weight above the 3rd percentile for age and sex per Centers for Disease Control and Prevention (CDC) World Health Organization (WHO) growth standards.
* Has received routine immunizations appropriate for age (as per national Center for Disease Control Advisory Committee on Immunization Practices [ACIP]). Note: COVID-19 vaccination will not be required unless fully licensed for this age group and ACIP-recommended. See study-specific Manual of Procedures for further guidance
* Is expected to be available for the duration of the study.
* If born to an HIV-infected woman, potential participant must have documentation of 2 negative HIV nucleic acid (RNA or DNA) test results from samples collected on different dates with both collected when greater than or equal to 4 weeks of age and at least one collected when greater than or equal to 16 weeks of age, and no positive HIV nucleic acid (RNA or DNA) test; or 2 negative HIV antibody tests, both from samples collected at greater than or equal to 24 weeks of age. If potential participant was breastfed by an HIV-infected woman, each of the sampling times noted above must be measured in weeks after the last exposure to breast milk, rather than weeks of age.

Exclusion Criteria:

* Prior laboratory-confirmed RSV infection.
* Known or suspected HIV infection or impairment of immunological functions.
* Receipt of immunosuppressive therapy, including any systemic, nasal, or inhaled corticosteroids within 28 days of enrollment. Note: Cutaneous (topical) steroid treatment is not an exclusion.
* Any receipt of bone marrow/solid organ transplant.
* Major congenital malformations (such as congenital cleft palate) or cytogenetic abnormalities.
* Previous enrollment in this trial, previous pediatric receipt of a licensed or investigational RSV vaccine, or previous maternal or pediatric receipt of or planned administration of any other anti-RSV product (such as ribavirin or RSV IG or RSV monoclonal antibody [mAb]) within 4 months of screening or planned administration of an anti-RSV product between screening and day 56 after enrollment.
* Any previous anaphylactic reaction.
* Any known hypersensitivity to any study product component.
* Heart disease. Note: Potential participants with cardiac abnormalities documented to be clinically insignificant and requiring no treatment may be enrolled.
* Lung disease, including any history of reactive airway disease or medically diagnosed wheezing.
* Member of a household that contains a person with chronic lung disease, including but not limited to chronic obstructive pulmonary disease (COPD), emphysema, or home oxygen use, reactive airway disease or asthma. Note: Asthma or reactive airway disease in a household member is not exclusionary unless the household member has taken oral steroids for asthma management in the past month and/or has been hospitalized for asthma in the past month.
* Member of a household that contains, or will contain, an infant who is less than 4 months of age at the enrollment date through Day 14.
* Member of a household that contains another child/other children who is/are enrolled or is/are scheduled to be enrolled in IMPAACT 2021 on a different date and has/have not completed the Day 56 visit in the same calendar year (i.e., all eligible children from the same household must be enrolled/receive study product on the same date or additional children in the household may be screened, enrolled, and randomized independently after other children in the household complete the Day 56 Visit).
* Member of a household that contains another child who is, or is scheduled to be, enrolled in another study evaluating an intranasal live-attenuated RSV vaccine, AND there has been or will be an overlap in residency during Day 0 to 14 of that other child's participation in the study.
* Member of a household that contains an immunocompromised individual, including, but not limited to:

  * a person who has been diagnosed with cancer and who has received chemotherapy within the 12 months prior to enrollment; or
  * a person living with a solid organ, cord blood, or bone marrow transplant.
* Shares a daycare room with infants less than 4 months of age, and parent/guardian is unable or unwilling to suspend daycare for 14 days following study product administration.
* Any of the following events at the time of enrollment:

  * fever (rectal temperature of greater than or equal to 100.4°F (38°C)), or
  * upper respiratory signs or symptoms (including but not limited to rhinorrhea, cough, or pharyngitis) or
  * nasal congestion significant enough to interfere with successful study product administration, or
  * otitis media.
  * Note: if participant is randomized and subsequently noted to have any of the above, study product administration must be deferred per the study protocol.
* Receipt of the following prior to enrollment (start counting backwards with '1' as the day of planned study product administration):

  * any inactivated vaccine or live-attenuated rotavirus vaccine within the 14 days prior, or
  * any live vaccine, other than rotavirus vaccine, within the 28 days prior, or
  * another investigational vaccine or investigational drug within 28 days prior. Note: if COVID-19 vaccine has EUA approval and ACIP recommendation for this age group, it is not considered investigational
* Scheduled administration of the following after planned study product administration (start counting with '1' as the day of planned study product administration):

  * inactivated vaccine or live-attenuated rotavirus vaccine within the 14 days after, or
  * any live vaccine other than rotavirus in the 28 days after, or
  * another investigational vaccine or investigational drug in the 56 days after. Note: if COVID-19 vaccine has EUA approval and ACIP recommendation for this age group, it is not considered investigational.
* Receipt of immunoglobulin, any antibody products, or any blood products within the past 6 months prior to enrollment
* Receipt of any of the following medications within 3 days prior to study enrollment:

  * systemic antibacterial, antiviral, antifungal, anti-parasitic, or antituberculous agents, whether for treatment or prophylaxis, or
  * intranasal medications, or
  * other prescription medication except as listed below
  * Permitted concomitant medications (prescription or non-prescription) include nutritional supplements, medications for gastroesophageal reflux, eye drops, and topical medications, including (but not limited to) cutaneous (topical) steroids, topical antibiotics, and topical antifungal agents.
* Born at less than 34 weeks gestation.
* Born between 34 weeks gestation and 36 weeks and 6 days gestation and less than 1 year of age at the time of enrollment.
* Current suspected or documented developmental disorder, delay, or other developmental problem.
* Any previous receipt of supplemental oxygen therapy in a home setting.
* Known or suspected SARS-CoV-2 exposure within the 14 days prior to enrollment. Note: known or suspected SARS-CoV-2 includes a known asymptomatic household member under quarantine for SARS-CoV-2 exposure but without a positive SARS-CoV-2 test.

Ages: 6 Months to 25 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 67 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Coleen Cunningham, MD, Study Chair — University of California, Irvine; Ruth Karron, MD, Study Chair — Center for Immunization Research (CIR), Johns Hopkins Bloomberg School of Public Health (JHSPH)
Locations (14):
- United States (14):
  - David Geffen School of Medicine at UCLA NICHD CRS, Los Angeles, California
  - University of California, UC San Diego CRS- Mother-Child-Adolescent HIV Program, San Diego, California
  - Univ. of Colorado Denver NICHD CRS, Aurora, Colorado
  - Emory University School of Medicine NICHD CRS, Atlanta, Georgia
  - Rush Univ. Cook County Hosp. Chicago NICHD CRS, Chicago, Illinois
  - Lurie Children's Hospital of Chicago (LCH) CRS, Chicago, Illinois
  - University of Maryland School of Medicine Center for Vaccine Development CRS, Baltimore, Maryland
  - The Children's Mercy Hospital CRS, Kansas City, Missouri
  - Center for Vaccine Development CRS, St Louis, Missouri
  - SUNY Stony Brook NICHD CRS, Stony Brook, New York
  - Jacobi Med. Ctr. Bronx NICHD CRS, The Bronx, New York
  - Duke Vaccine and Trials Unit CRS, Durham, North Carolina
  - Gamble Center for Clinical Studies CRS, Cincinnati, Ohio
  - Baylor College of Medicine/ Texas Children's Hospital NICHD CRS, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the International Maternal Pediatric Adolescent AIDS Clinical Trial (IMPAACT) Network by NIH.
Access Criteria: * With whom?
    * Researchers who provide a methodologically sound proposal for use of the data that is approved by the IMPAACT Network.
  * For what types of analyses?
    * To achieve aims in the proposal approved by the IMPAACT Network.
  * By what mechanism will data be made available?
    * Researchers may submit a request for access to data using the IMPAACT "Data Request" form at: https://www.impaactnetwork.org/studies/submit-research-proposals. Researchers of approved proposals will need to sign an IMPAACT Data Use Agreement before receiving the data.
URL: https://www.impaactnetwork.org/studies/submit-research-proposal

REFERENCES:
- See also: The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), corrected Version 2.1 July 2017 — https://rsc.niaid.nih.gov/clinical-research-sites/daids-adverse-event-grading-tables
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — https://rsc.niaid.nih.gov/clinical-research-sites/manual-expedited-reporting-adverse-events-daids

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RSV ΔNS2/Δ1313/I1314L Vaccine | RSV 6120/ΔNS2/1030s Vaccine | RSV 276 Vaccine | Placebo
Started | 20 | 20 | 7 | 20
Completed | 18 | 19 | 7 | 19
Not Completed | 2 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Moved | 1 | 0 | 0 | 1
Not completed — Not Able to Get to Clinic | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RSV ΔNS2/Δ1313/I1314L Vaccine | RSV 6120/ΔNS2/1030s Vaccine | RSV 276 Vaccine | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 7 | 20 | 67
Age, Continuous [Median (Inter-Quartile Range); unit: Months] | 12.4 [10.0 to 19.5] | 14.6 [8.2 to 17.3] | 16.5 [9.1 to 21.6] | 12.3 [8.1 to 15.2] | 13.3 [8.6 to 18.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 4 | 9 | 32
  Male | 12 | 9 | 3 | 11 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 3 | 7 | 16
  Not Hispanic or Latino | 17 | 17 | 4 | 13 | 51
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 5 | 1 | 7 | 19
  White | 11 | 14 | 6 | 11 | 42
  More than one race | 1 | 1 | 0 | 0 | 2
  Unknown or Not Reported | 1 | 0 | 0 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 7 | 20 | 67
HIV Exposure (from maternal HIV status) [Count of Participants; unit: Participants]
  Not HIV Exposed | 12 | 15 | 6 | 10 | 43
  HIV Exposed | 8 | 5 | 1 | 10 | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage With Grade 1 or Higher Solicited Adverse Events (AEs)
Description: Solicited adverse events include fever, otitis media, upper respiratory illness (URI), and lower respiratory illness (LRI) and are graded following a protocol-defined grading system. Adverse events were graded on a scale from 1-5: 1=mild, 2=moderate, 3=severe, 4=life-threatening, 5=death. All solicited AEs with at least mild severity were included. Percentage with 95% exact confidence intervals using the Clopper-Pearson method were calculated.
Time Frame: Day 0 through Day 28
Population: All participants who received study product
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RSV ΔNS2/Δ1313/I1314L Vaccine | RSV 6120/ΔNS2/1030s Vaccine | RSV 276 Vaccine | Placebo
Number analyzed (Participants) | 20 | 20 | 7 | 20
percentage of participants | 55 [32 to 77] | 40 [19 to 64] | 71 [29 to 96] | 55 [32 to 77]
Statistical Analysis 1: Comparison: RSV ΔNS2/Δ1313/I1314L Vaccine vs Placebo; Test type: Superiority; p > 0.99, Fisher Exact — Statistical significance level of 0.05 was used. No adjustment for multiple comparisons; Difference in proportions = 0, 95% CI 2-sided [-32 to 32] — Comparison was vaccine arm - placebo
Statistical Analysis 2: Comparison: RSV 6120/ΔNS2/1030s Vaccine vs Placebo; Test type: Superiority; p = 0.53, Fisher Exact — Statistical significance level of 0.05 used. No adjustments made for multiple comparisons; Difference in proportions = -15, 95% CI 2-sided [-46 to 18] — Comparison was vaccine arm - placebo
Statistical Analysis 3: Comparison: RSV 276 Vaccine vs Placebo; Test type: Superiority; p = 0.66, Fisher Exact — Statistical significance level of 0.05 was used. No adjustments made for multiple comparisons; Difference in proportions = 16, 95% CI 2-sided [-29 to 52] — Comparison was vaccine arm - placebo

2. Primary Outcome: Percentage With Grade 2 or Higher Lower Respiratory Illnesses (LRIs)
Description: LRIs graded following a protocol-defined grading system. Adverse events were graded on a scale from 1-5: 1=mild, 2=moderate, 3=severe, 4=life-threatening, 5=death. All solicited LRIs with at least moderate severity were included. Percentage with 95% exact confidence intervals using the Clopper-Pearson method were calculated.
Time Frame: Day 0 through Day 28
Population: All participants who received study product
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RSV ΔNS2/Δ1313/I1314L Vaccine | RSV 6120/ΔNS2/1030s Vaccine | RSV 276 Vaccine | Placebo
Number analyzed (Participants) | 20 | 20 | 7 | 20
percentage of participants | 5 [0 to 25] | 0 [0 to 17] | 0 [0 to 41] | 5 [0 to 25]
Statistical Analysis 1: Comparison: RSV ΔNS2/Δ1313/I1314L Vaccine vs Placebo; Test type: Superiority; p > 0.99, Fisher Exact — Statistical significance level of 0.05 was used. No adjustments made for multiple comparisons; Difference in proportions = 0, 95% CI 2-sided [-20 to 20] — Comparison was vaccine arm - placebo
Statistical Analysis 2: Comparison: RSV 6120/ΔNS2/1030s Vaccine vs Placebo; Test type: Superiority; p > 0.99, Fisher Exact — Statistical significance level of 0.05 was used. No adjustments made for multiple comparisons; Difference in proportions = -5, 95% CI 2-sided [-25 to 13] — Comparison was vaccine arm - placebo
Statistical Analysis 3: Comparison: RSV 276 Vaccine vs Placebo; Test type: Superiority; p > 0.99, Fisher Exact — Statistical significance level of 0.05 was used. No adjustments made for multiple comparisons; Difference in proportions = -5, 95% CI 2-sided [-26 to 34] — Comparison was vaccine arm - placebo

3. Primary Outcome: Percentage With Serious AEs
Description: Serious adverse events are defined according to Version 2.0 of the DAIDS EAE Manual. A serious event is one that requires or lengthens hospitalization, that is life-threatening, that results in death, that results in a significant disability, or that is a congenital anomaly or birth defect. Percentage with 95% exact confidence intervals using the Clopper-Pearson method were calculated.
Time Frame: Day 0 through Day 56
Population: All participants who received study product
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RSV ΔNS2/Δ1313/I1314L Vaccine | RSV 6120/ΔNS2/1030s Vaccine | RSV 276 Vaccine | Placebo
Number analyzed (Participants) | 20 | 20 | 7 | 20
percentage of participants | 0 [0 to 17] | 0 [0 to 17] | 0 [0 to 41] | 0 [0 to 17]
Statistical Analysis 1: Comparison: RSV ΔNS2/Δ1313/I1314L Vaccine vs Placebo; Test type: Superiority; p > 0.99, Fisher Exact — Statistical significance level of 0.05 was used. No adjustments made for multiple comparisons; Difference in proportions = 0, 95% CI 2-sided [-18 to 18] — Comparison was vaccine arm - placebo
Statistical Analysis 2: Comparison: RSV 6120/ΔNS2/1030s Vaccine vs Placebo; Test type: Superiority; p > 0.99, Fisher Exact — Statistical significance level of 0.05 was used. No adjustments made for multiple comparisons; Difference in proportions = 0, 95% CI 2-sided [-18 to 18] — Comparison was vaccine arm - placebo
Statistical Analysis 3: Comparison: RSV 276 Vaccine vs Placebo; Test type: Superiority; p > 0.99, Fisher Exact — Statistical significance level of 0.05 was used. No adjustments made for multiple comparisons; Difference in proportions = 0, 95% CI 2-sided [-17 to 41] — Comparison was vaccine arm - placebo

4. Primary Outcome: Percentage With a Greater Than or Equal to 4-fold Rise in Serum RSV-neutralizing Antibody Titer
Description: Antibody responses were defined as a greater than or equal to 4-fold increase in titer in paired specimens, between pre-study product administration and Day 56 time points. Percentage with 95% exact confidence intervals (CIs) using the Clopper-Pearson method were calculated. The upper limit of the CI was compared to an a priori limit of 70%. An upper limit above 70% was considered a good vaccine candidate.
Time Frame: Measured at pre-study product administration (screening) through Day 56
Population: Participants with samples available at baseline and Day 56, with Day 56 Visit in the protocol-defined visit window, and one participant randomly selected from households with more than one child enrolled on the same date
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RSV ΔNS2/Δ1313/I1314L Vaccine | RSV 6120/ΔNS2/1030s Vaccine | RSV 276 Vaccine | Placebo
Number analyzed (Participants) | 17 | 17 | 7 | 20
percentage of participants | 76 [50 to 93] | 71 [44 to 90] | 71 [29 to 96] | 15 [3 to 38]
Statistical Analysis 1: Comparison: RSV ΔNS2/Δ1313/I1314L Vaccine vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — Statistical significance level of 0.05 was used. No adjustment for multiple comparisons; Difference in proportions = 61, 95% CI 2-sided [27 to 83] — Comparison was vaccine arm - placebo
Statistical Analysis 2: Comparison: RSV 6120/ΔNS2/1030s Vaccine vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact; Statistical significance level of 0.05 was used. No adjustments made for multiple comparisons; Difference in proportions = 56, 95% CI 2-sided [22 to 79] — Comparison was vaccine arm - placebo
Statistical Analysis 3: Comparison: RSV 276 Vaccine vs Placebo; Test type: Superiority; p = 0.011, Fisher Exact; Statistical significance level of 0.05 was used. No adjustments were made for multiple comparisons; Difference in proportions = 56, 95% CI 2-sided [9 to 86] — Comparison was vaccine arm - placebo
Statistical Analysis 4: Comparison: RSV ΔNS2/Δ1313/I1314L Vaccine vs RSV 6120/ΔNS2/1030s Vaccine; Test type: Superiority; p > 0.99, Fisher Exact — Statistical significance level of 0.05 was used. No adjustments made for multiple comparisons; Difference in proportions = 6, 95% CI 2-sided [-25 to 36] — Comparison was RSV ΔNS2/Δ1313/I1314L Vaccine - RSV 6120/ΔNS2/1030s Vaccine
Statistical Analysis 5: Comparison: RSV ΔNS2/Δ1313/I1314L Vaccine vs RSV 276 Vaccine; Test type: Superiority; p > 0.99, Fisher Exact — Statistical significance level of 0.05 was used. No adjustments made for multiple comparisons; Difference in proportions = 5, 95% CI 2-sided [-31 to 48] — Comparison was RSV ΔNS2/Δ1313/I1314L Vaccine - RSV 276 Vaccine
Statistical Analysis 6: Comparison: RSV 6120/ΔNS2/1030s Vaccine vs RSV 276 Vaccine; Test type: Superiority; p > 0.99, Fisher Exact — Statistical significance level of 0.05 was used. No adjustments made for multiple comparisons; Difference in proportions = -1, 95% CI 2-sided [-38 to 44] — Comparison was RSV 6120/ΔNS2/1030s Vaccine - RSV 276 Vaccine

5. Secondary Outcome: Percentage With a Greater Than or Equal to 4-fold Rise in Serum RSV F Immunoglobulin G (IgG)
Description: RSV F IgG responses were defined as a greater than or equal to 4-fold increase in titer in paired specimens, between pre-study product administration and Day 56 time points. Percentage with 95% exact CIs using the Clopper-Pearson method were calculated. The upper limit of the CI was compared to an a priori level of 70%. An upper limit above 70% was considered a good vaccine candidate.
Time Frame: Measured at pre-study product administration (screening) and Day 56
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RSV ΔNS2/Δ1313/I1314L Vaccine | RSV 6120/ΔNS2/1030s Vaccine | RSV 276 Vaccine | Placebo
Number analyzed (Participants) | 17 | 17 | 7 | 20
percentage of participants | 88 [64 to 99] | 76 [50 to 93] | 100 [59 to 100] | 15 [3 to 38]
Statistical Analysis 1: Comparison: RSV ΔNS2/Δ1313/I1314L Vaccine vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — Statistical significance level of 0.05 was used. No adjustments made for multiple comparisons; Difference in proportions = 73, 95% CI 2-sided [44 to 91] — Comparison was vaccine arm - placebo
Statistical Analysis 2: Comparison: RSV 6120/ΔNS2/1030s Vaccine vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — Statistical significance level of 0.05 was used. No adjustments made for multiple comparisons; Difference in proportions = 61, 95% CI 2-sided [27 to 83] — Comparison was vaccine arm - placebo
Statistical Analysis 3: Comparison: RSV 276 Vaccine vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — Statistical significance level of 0.05 was used. No adjustments made for multiple comparisons; Difference in proportions = 85, 95% CI 2-sided [42 to 97] — Comparison was vaccine arm - placebo
Statistical Analysis 4: Comparison: RSV ΔNS2/Δ1313/I1314L Vaccine vs RSV 6120/ΔNS2/1030s Vaccine; Test type: Superiority; p = 0.66, Fisher Exact — Statistical significance level of 0.05 was used. No adjustments made for multiple comparisons; Difference in proportions = 12, 95% CI 2-sided [-17 to 40] — Comparison was RSV ΔNS2/Δ1313/I1314L Vaccine - RSV 6120/ΔNS2/1030s Vaccine
Statistical Analysis 5: Comparison: RSV ΔNS2/Δ1313/I1314L Vaccine vs RSV 276 Vaccine; Test type: Superiority; p > 0.99, Fisher Exact — Statistical significance level of 0.05 was used. No adjustments made for multiple comparisons; Difference in proportions = -12, 95% CI 2-sided [-36 to 30] — Comparison was RSV ΔNS2/Δ1313/I1314L Vaccine - RSV 276 Vaccine
Statistical Analysis 6: Comparison: RSV 6120/ΔNS2/1030s Vaccine vs RSV 276 Vaccine; Test type: Superiority; p = 0.28, Fisher Exact — Statistical significance level of 0.05 was used. No adjustments made for multiple comparisons; Difference in proportions = -24, 95% CI 2-sided [-50 to 20] — Comparison was RSV 6120/ΔNS2/1030s Vaccine - RSV 276 Vaccine

6. Secondary Outcome: Titer of Serum RSV F IgG
Description: Serum F IgG antibodies were assessed by Enzyme-linked Immunosorbent Assay (ELISA). Titers below the limit of detection (1:50) were assigned a value equal to half the corresponding limit of detection (1:25) and evaluated as reciprocals of the titer (log2).
Time Frame: Measured at the Day 56 Visit
Population: Participants with a Day 56 sample available, with the Day 56 visit in the protocol-defined visit window, and one participant randomly selected from households with more than one child enrolled on the same date
Measure: Median (Inter-Quartile Range); unit: log 2 titers
Arm/Group | RSV ΔNS2/Δ1313/I1314L Vaccine | RSV 6120/ΔNS2/1030s Vaccine | RSV 276 Vaccine | Placebo
Number analyzed (Participants) | 17 | 17 | 7 | 20
log 2 titers | 12.0 [11.0 to 12.5] | 12.0 [10.7 to 12.4] | 14.3 [12.6 to 15.5] | 4.6 [4.6 to 8.4]
Statistical Analysis 1: Comparison: RSV ΔNS2/Δ1313/I1314L Vaccine vs Placebo; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — Statistical significance level of 0.05 was used. No adjustments made for multiple comparisons
Statistical Analysis 2: Comparison: RSV 6120/ΔNS2/1030s Vaccine vs Placebo; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — Statistical significance level of 0.05 was used. No adjustments made for multiple comparisons
Statistical Analysis 3: Comparison: RSV 276 Vaccine vs Placebo; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — Statistical significance of 0.05 was used. No adjustments made for multiple comparisons
Statistical Analysis 4: Comparison: RSV ΔNS2/Δ1313/I1314L Vaccine vs RSV 6120/ΔNS2/1030s Vaccine; Test type: Superiority; p = 0.95, Wilcoxon (Mann-Whitney) — Statistical significance level of 0.05 was used. No adjustments made for multiple comparisons
Statistical Analysis 5: Comparison: RSV ΔNS2/Δ1313/I1314L Vaccine vs RSV 276 Vaccine; Test type: Superiority; p = 0.12, Wilcoxon (Mann-Whitney) — Statistical significance level of 0.05 was used. No adjustments made for multiple comparisons
Statistical Analysis 6: Comparison: RSV 6120/ΔNS2/1030s Vaccine vs RSV 276 Vaccine; Test type: Superiority; p = 0.033, Wilcoxon (Mann-Whitney) — Statistical significance level of 0.05 was used. No adjustments made for multiple comparisons

7. Secondary Outcome: Titer of Serum RSV-neutralizing Antibodies
Description: Serum RSV-neutralizing antibody titers were assessed by RSV-plaque reduction neutralization titer (RSV-PRNT) assay. Titers below the limit of detection (1:10) were assigned a value equal to half the corresponding limit of detection (1:5) and evaluated as reciprocals of the titer (log2).
Time Frame: Measured at the Day 56 Visit
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: log 2 titers
Arm/Group | RSV ΔNS2/Δ1313/I1314L Vaccine | RSV 6120/ΔNS2/1030s Vaccine | RSV 276 Vaccine | Placebo
Number analyzed (Participants) | 17 | 17 | 7 | 20
log 2 titers | 6.2 [4.3 to 7.3] | 5.1 [4.5 to 6.3] | 7.7 [6.5 to 9.3] | 2.3 [2.3 to 3.4]
Statistical Analysis 1: Comparison: RSV ΔNS2/Δ1313/I1314L Vaccine vs Placebo; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — Statistical significance level of 0.05 was used. No adjustments made for multiple comparisons
Statistical Analysis 2: Comparison: RSV 6120/ΔNS2/1030s Vaccine vs Placebo; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — Statistical significance level of 0.05 was used. No adjustments made for multiple comparisons
Statistical Analysis 3: Comparison: RSV 276 Vaccine vs Placebo; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — Statistical significance level of 0.05 was used. No adjustments made for multiple comparisons
Statistical Analysis 4: Comparison: RSV ΔNS2/Δ1313/I1314L Vaccine vs RSV 6120/ΔNS2/1030s Vaccine; Test type: Superiority; p = 0.39, Wilcoxon (Mann-Whitney) — Statistical significance level of 0.05 was used. No adjustments made for multiple comparisons
Statistical Analysis 5: Comparison: RSV ΔNS2/Δ1313/I1314L Vaccine vs RSV 276 Vaccine; Test type: Superiority; p = 0.15, Wilcoxon (Mann-Whitney) — Statistical significance level of 0.05 was used. No adjustments made for multiple comparisons
Statistical Analysis 6: Comparison: RSV 6120/ΔNS2/1030s Vaccine vs RSV 276 Vaccine; Test type: Superiority; p = 0.049, Wilcoxon (Mann-Whitney) — Statistical significance level of 0.05 was used. No adjustments made for multiple comparisons

8. Secondary Outcome: Percentage With RSV-associated Medically Attended Acute Respiratory Illness (RSV-MAARI)
Description: The percentage and 95% exact Clopper-Pearson CI of participants who had RSV-associated, symptomatic, medically attended respiratory and febrile illness (MAARI) among those who had indicators of natural infection with wt RSV were presented. Natural infection with wild type (wt) RSV during the RSV season surveillance period was defined as having either RSV detected in nasal samples collected during illness visits for MAARI events or through site reporting. RSV-associated upper respiratory tract illness, lower respiratory tract illness, otitis media, or fever were graded following a protocol-defined grading system.
Time Frame: Measured through the last day of the RSV season, which will occur between 5 and 15 months after study entry, depending on when the participant enrolls in the study
Population: Participants with follow up during an RSV season
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RSV ΔNS2/Δ1313/I1314L Vaccine | RSV 6120/ΔNS2/1030s Vaccine | RSV 276 Vaccine | Placebo
Number analyzed (Participants) | 19 | 20 | 7 | 20
percentage of participants | 11 [1 to 33] | 15 [3 to 38] | 0 [0 to 41] | 5 [0 to 25]

9. Secondary Outcome: Maximum Grade (if More Than One Illness Within a Participant) of RSV-MAARI
Description: The number of participants who had RSV-MAARI among those who had indicators of natural infection with wt RSV were presented. Natural infection with wt RSV during the RSV season surveillance period was defined as having either RSV detected in nasal samples collected during illness visits for MAARI events or through site reporting. A participant was only counted once in the line corresponding to the highest grade MAARI event they experienced. These events were graded following a protocol-defined grading system. Adverse events were graded on a scale from 1-5: 1=mild, 2=moderate, 3=severe, 4=life-threatening, 5=death.
Time Frame: as for outcome 8
Population: Participants with follow up during an RSV season
Measure: Count of Participants; unit: Participants
Arm/Group | RSV ΔNS2/Δ1313/I1314L Vaccine | RSV 6120/ΔNS2/1030s Vaccine | RSV 276 Vaccine | Placebo
Number analyzed (Participants) | 19 | 20 | 7 | 20
Participants
  No RSV-MAARI | 17 | 17 | 7 | 19
  Grade 1 | 0 | 1 | 0 | 1
  Grade 2 | 2 | 2 | 0 | 0

10. Secondary Outcome: Percentage With RSV-associated Medically Attended Acute Lower Respiratory Illness (RSV-MAALRI)
Description: The percentage and 95% exact Clopper-Pearson CI of participants who had RSV-associated, symptomatic, medically attended acute lower respiratory tract illness (MAALRI) among those who had indicators of natural infection with wt RSV were presented. Natural infection with wt RSV during the RSV season surveillance period was defined as having either RSV detected in nasal samples collected during illness visits for MAALRI events or through site reporting. RSV-associated lower respiratory tract illness graded following a protocol-defined grading system.
Time Frame: as for outcome 8
Population: Participants will follow up during an RSV season
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RSV ΔNS2/Δ1313/I1314L Vaccine | RSV 6120/ΔNS2/1030s Vaccine | RSV 276 Vaccine | Placebo
Number analyzed (Participants) | 19 | 20 | 7 | 20
percentage of participants | 5 [0 to 26] | 0 [0 to 17] | 0 [0 to 41] | 0 [0 to 17]

11. Secondary Outcome: Maximum Grade (if More Than One Illness Within a Participant) of RSV-MAALRI
Description: The number of participants who had RSV-MAALRI among those who had indicators of natural infection with wt RSV were presented. Natural infection with wt RSV during the RSV season surveillance period was defined as having either RSV detected in nasal samples collected during illness visits for MAALRI events or through site reporting. A participant was only counted once in the line corresponding to the highest grade MAALRI event they experienced. These events were graded following a protocol-defined grading system. Adverse events were graded on a scale from 1-5: 1=mild, 2=moderate, 3=severe, 4=life-threatening, 5=death.
Time Frame: as for outcome 8
Population: Participants with follow up during an RSV season
Measure: Count of Participants; unit: Participants
Arm/Group | RSV ΔNS2/Δ1313/I1314L Vaccine | RSV 6120/ΔNS2/1030s Vaccine | RSV 276 Vaccine | Placebo
Number analyzed (Participants) | 19 | 20 | 7 | 20
Participants
  No RSV-MAALRI | 18 | 20 | 7 | 20
  Grade 1 | 0 | 0 | 0 | 0
  Grade 2 | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 5 to 12 months depending on when a participant enrolled and how close the enrollment was to the start of RSV season
Description: All adverse events collected through Day 28. All serious AEs collected through Day 56. From Day 56 to RSV Season only serious and unexpected suspected adverse reactions (SUSARs) collected. During RSV season only medically attended fevers, LRIs, URIs, and otitis media, as well as all serious AEs collected. At the Post-RSV season visit, only SUSARs and grade 3 or higher AEs related to visit procedures collected.
Arm/Group | RSV ΔNS2/Δ1313/I1314L Vaccine | RSV 6120/ΔNS2/1030s Vaccine | RSV 276 Vaccine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/7 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/7 | 0/20
Other Adverse Events (participants affected / at risk) | 14/20 | 11/20 | 6/7 | 13/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RSV ΔNS2/Δ1313/I1314L Vaccine (N=20) | RSV 6120/ΔNS2/1030s Vaccine (N=20) | RSV 276 Vaccine (N=7) | Placebo (N=20)
Eye discharge (Eye disorders) | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 1 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Lip swelling (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Teething (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Developmental delay (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 4 | 5 | 5 | 8
Swelling face (General disorders) | 1 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Adenovirus infection (Infections and infestations) | 1 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 1 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 1
Conjunctivitis viral (Infections and infestations) | 0 | 0 | 0 | 1
Croup infectious (Infections and infestations) | 1 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 1 | 0 | 0 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 3 | 3 | 4 | 2
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 1
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 6 | 5 | 2 | 2
Cardiac murmur (Investigations) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0
Infant irritability (Nervous system disorders) | 2 | 2 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 2 | 6
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 10 | 10 | 5 | 9
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Eczema infantile (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The study closed to enrollment prior to fully accruing. As a result, outcomes were estimated with less precision than originally planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol and Informed Consent Form: Protocol Version 3.0 (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/85/NCT03916185/Prot_ICF_000.pdf
  • Study Protocol: Clarification Memo 1 (2023-01-18): https://cdn.clinicaltrials.gov/large-docs/85/NCT03916185/Prot_001.pdf
  • Study Protocol: Letter of Amendment 1 (2023-09-25): https://cdn.clinicaltrials.gov/large-docs/85/NCT03916185/Prot_002.pdf
  • Statistical Analysis Plan (2023-11-07): https://cdn.clinicaltrials.gov/large-docs/85/NCT03916185/SAP_003.pdf